CLINICAL TRIAL: NCT03226834
Title: Comparison of Musicotherapy Sessions Using Patient Play-list Versus U Sequence Music Care Medical Device on Pre-operative Anxiety in Women Undergoing Gynecological Surgery: a Randomized-control Study
Brief Title: Efficiency of Favourite Versus Predetermined Musical Sequence on Gynecology Pre-operative Anxiety
Acronym: MUANX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016/CHU/04
Record Dates: First submitted 2017-07-18; First posted 2017-07-24 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Surgery; Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: control randomized, single blind, monocentric
Who Masked: Care Provider, Investigator
Masking Description: blindness concerns medical staff: nurses in charge of the blood parameters measurements as well as anxiety evaluation are not informed of the allocation of the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUSIC CARE (Active Comparator): Listening for 20 min of one of the music style U sequences proposed by the medical device MUSIC CARE
  Interventions: Device: MUSIC CARE
- PERSONAL PLAY-LIST (Experimental): Listening for 20 min of patient's play-list
  Interventions: Other: PERSONAL PLAY-LIST

INTERVENTIONS:
Device: MUSIC CARE — Musicotherapy session using one of the U musical sequences of MUSIC CARE among the preselected music styles
  Other Names: Music Care U sequence
  Arms: MUSIC CARE
Other: PERSONAL PLAY-LIST — Musicotherapy session using the patient's play-list composed by the patient with her favourite songs
  Other Names: Patient's paly-list
  Arms: PERSONAL PLAY-LIST

SUMMARY:
Anxiety is a psychologic and physiological state that could be characterized by somatic, emotional, cognitive and behavioral components. Surgery, as well as waiting for surgery is an anxiogenic situation encountered by 60 à 80 % of the patients. High levels of anxiety lead to negative physiological signs that slow down healing, lowers imune response and increases post-surgery infection. Anxiety also increases pain and post-surgery morbi-mortality. Drug-induced sedation is frequently recommended to lower anxiety. The anxiolytic effect of alternative treatment such as musicotherapy has been demonstrated in several randomized control trials. Nevertheless, most of these studies have investigated the effect of musicotherapy in groups with our without musical listening.

In the present study, investigators assume that a personal musical sequence composed by favourite songs of the patients could have beneficial effect on presurgical anxiety than selective sequence of the medical device MUSIC CARE.

In this study, the anxiolytic effect of predefined U musical sequences that alternate slow and faster music tracks (medical device MUSIC CARE) are compared to patient's play-list, in women with planned gynecological surgery.

DETAILED DESCRIPTION:
Patients are randomly allocated in two groups:

* control group: patients are asked to choose one of the U sequence among the preselected music style proposed by the medical device MUSIC CARE
* test group: patients are asked to prepare their own play-list containing their favourite songs

Anxiety is assessed before and after a 20 min-musicotherapy session by using the State-Trait Anxiety Inventory (STAI) for anxiogenic situation.

Other parameters are measured such as blood pressure, cardiac frequency, level of pain after surgery, care stay duration, potent post-surgery complications.

ELIGIBILITY:
Inclusion Criteria:

* with planed gynecologic surgery
* without anxiolytic medication
* able to prepare their own play-list
* signed inform consent

Exclusion Criteria:

* hearing disorder
* dementia or psychiatric disorder
* neurologic disorder

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-09-22 (Actual)

PRIMARY OUTCOMES:
Situation anxiety measurement | Change from baseline anxiety at 20 minutes musical listening
  Pre-operative anxiety is assessed by the STAY-situation questionnaire

SECONDARY OUTCOMES:
Blood pressure | Change from baseline blood pressure at 20 minutes musical listening
  Measurement of blood pressure
Post-operative pain | Up to one hour after surgery recovery
  Pain is assessed after surgery recovery using Visual Analogic Scale
Care stay duration | At study completion, an average of 3 days
  Hospital stay is assessed by the number of days
Post-operative complications | Through study completion, an average of 3 days
  All post-operative complications are recorded
Heart rate | Change from baseline heart at 20 minutes musical listening
  Measurement of heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Malik Boukerrou, MD, Principal Investigator — Centre Hpospitalier Universitaire de La REUNION
Locations (1):
- Chu Reunion Island, Saint-Pierre, Reunion Island, Reunion

REFERENCES:
- [Derived] Reynaud D, Bouscaren N, Lenclume V, Boukerrou M. Comparing the effects of self-selected MUsic versus predetermined music on patient ANXiety prior to gynaecological surgery: the MUANX randomized controlled trial. Trials. 2021 Aug 13;22(1):535. doi: 10.1186/s13063-021-05511-2. PMID 34389022
- [Derived] Petot T, Bouscaren N, Maillard O, Huiart L, Boukerrou M, Reynaud D. Comparing the effects of self-selected music versus predetermined music on patient anxiety prior to gynaecological surgery: a study protocol for a randomised controlled trial. Trials. 2019 Jan 7;20(1):20. doi: 10.1186/s13063-018-3093-6. PMID 30616674